CLINICAL TRIAL: NCT03299946
Title: Feasibility and Efficacy of Neoadjuvant Cabozantinib Plus Nivolumab (CaboNivo) Followed by Definitive Resection for Patients With Locally Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Exelixis (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J17136; IRB00149350 (Other: Johns Hopkins University)
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Hepatocellular Carcinoma
Keywords: Nivolumab; Cabozantinib; Neoadjuvant; Immunotherapy; Liver Cancer; Borderline Resectable; Advance Resectable; Neoplasms; Hepatocellular Carcinoma; HCC; Resection
MeSH Terms: conditions — Liver Neoplasms; Neoplasms; Carcinoma, Hepatocellular | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Cabozantinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib (40mg) will be taken by mouth daily for 8 weeks.
  Other Names: XL184
Drug: Nivolumab — Nivolumab 240mg intravenously every 2 weeks (days 14, 28, 42, and 56 for a total of four doses), in combination with Cabozantinib 40mg by mouth daily for 8 weeks.
  Other Names: OPDIVO, BMS 936558, MDX-1106, ONO-4538

SUMMARY:
The proposed study is an open-label, single institution, single arm phase 1b study of neoadjuvant cabozantinib plus nivolumab in patients with locally advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Must have locally advanced/borderline resectable hepatocellular carcinoma.
2. Must have measurable disease.
3. Age ≥18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
6. Patients must have adequate liver remnant and function.
7. Antiviral therapy per local standard of care for hepatitis B.
8. Woman of child bearing potential must have a negative pregnancy test.
9. Must use acceptable form of birth control while on study.
10. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed HCC.
2. Chemotherapy, radiotherapy, investigational therapy, or surgery less than 6 months prior to trial registration.
3. Concomitant Anticoagulation therapy.
4. Any GI or pulmonary risks of bleeding.
5. History of HIV Infection.
6. Active co-infection with hepatitis B and hepatitis C.
7. Active co-infection with hepatitis B and hepatitis D.
8. Has a diagnosis of immunodeficiency, or is receiving systemic steroid therapy.
9. History of any autoimmune disease requiring systemic treatment within the past 2 years. Any patient bearing an allograft is not eligible.
10. Any additional malignancies with treatment or life-limiting cancers. Superficial bladder cancer, non-melanoma skin cancers, or low grade prostate cancer not requiring therapy would not exclude participation in this trial.
11. Uncontrolled intercurrent illness.
12. Corrected QT interval calculated by the Fridericia formula.
13. Uncontrolled high blood pressure.
14. Are pregnant or breastfeeding.
15. Any gastrointestinal (GI) disorders.
16. Any certain study-specified heart conditions 6 months prior to enrollment.
17. Major surgery within 2 months before enrollment.
18. Have any evidence of moderate or severe ascites.
19. Any untreated or incompletely treated varices with bleeding or high-risk bleeding.
20. Inability to swallow intact tablets.
21. Known or suspected hypersensitivity to study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events in participants of neoadjuvant cabozantinib plus nivolumab. | 4 years
Number of patients who complete pre-op treatment and proceed to surgery. | 4 years

SECONDARY OUTCOMES:
Percentage of participants who obtain R0 resection. | 4 years
Percentage of participants who obtain a pathologic complete response (CR). | 4 years
Percentage of participants who obtain a major pathologic responses (MPR) | 4 years
Objective response rate (ORR) | 4 years
Median Overall Survival (OS) | 5 years
Disease free survival (DFS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laheru, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang S, Yuan L, Danilova L, Mo G, Zhu Q, Deshpande A, Bell ATF, Elisseeff J, Popel AS, Anders RA, Jaffee EM, Yarchoan M, Fertig EJ, Kagohara LT. Spatial transcriptomics analysis of neoadjuvant cabozantinib and nivolumab in advanced hepatocellular carcinoma identifies independent mechanisms of resistance and recurrence. Genome Med. 2023 Sep 18;15(1):72. doi: 10.1186/s13073-023-01218-y. PMID 37723590
- [Derived] Ho WJ, Zhu Q, Durham J, Popovic A, Xavier S, Leatherman J, Mohan A, Mo G, Zhang S, Gross N, Charmsaz S, Lin D, Quong D, Wilt B, Kamel IR, Weiss M, Philosophe B, Burkhart R, Burns WR, Shubert C, Ejaz A, He J, Deshpande A, Danilova L, Stein-O'Brien G, Sugar EA, Laheru DA, Anders RA, Fertig EJ, Jaffee EM, Yarchoan M. Neoadjuvant Cabozantinib and Nivolumab Converts Locally Advanced HCC into Resectable Disease with Enhanced Antitumor Immunity. Nat Cancer. 2021 Sep;2(9):891-903. doi: 10.1038/s43018-021-00234-4. Epub 2021 Jul 29. PMID 34796337